CLINICAL TRIAL: NCT06866613
Title: Randomized, Controlled, Double-blind, Multi-center Trial to Evaluate the Efficacy and Safety of an Esflurbiprofen Topical System (EFTS) vs. Placebo in the Local Symptomatic and Short-term Treatment of Pain in Ankle Sprains.
Brief Title: Phase III Trial to Evaluate the Efficacy and Safety in Patients With Ankle Sprains.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teikoku Seiyaku Co., Ltd. (Industry)
Collaborators: CRM Biometrics GmbH (Industry); SocraTec R&D GmbH (Other); SocraMetrics GmbH (Industry); HWI pharma services GmbH (Industry); Clinsearch GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TK-254RX-0301; 2024-513063-45-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-10; First posted 2025-03-10 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-04

CONDITIONS: Ankle Sprains
Keywords: Blunt trauma; Soft tissue injuries; sports injuries; NSAIDs; topical patch
MeSH Terms: conditions — Ankle Injuries; Wounds, Nonpenetrating; Soft Tissue Injuries; Athletic Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TK-254RX (Experimental): Esflurbiprofen Topical System 165 mg Esflurbiprofen
  Interventions: Drug: Esflurbiprofen Topical System (EFTS)
- Placebo patch (Placebo Comparator): Placebo patch does not contain active ingredients but it cannot be distinguished in terms of appearance, consistency, odor, and dosage form
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Esflurbiprofen Topical System (EFTS) — One EFTS is applied to the injured area over consecutive 7 days
  Arms: TK-254RX
Drug: Placebo Patch — One placebo patch is applied to the injured area over consecutive 7 days
  Arms: Placebo patch

SUMMARY:
This study is a multi-center, double-blind, randomized controlled trial to evaluate the efficacy and safety of EFTS vs. placebo in patients with ankle sprains. The primary objective of this study is to demonstrate that the EFTS is superior in pain reduction compared to a matching placebo in patients with ankle sprains.

The secondary objective is to evaluate tolerability, local tolerability, and adhesion of EFTS vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

* acute ankle sprains Grade I
* location of injury such that pain-on-movement (POM) is elicited on active standardized movement
* enrollment within 6 hours of the injury
* baseline VAS score for POM of injured extremity > 50 mm on a 100 mm VAS
* adult male or female patients
* age 18 to 64 years (including)
* having given written informed consent
* satisfactory health as determined by the Investigator based on medical history and physical examination.

Exclusion Criteria:

* significant concomitant injury in association with the index soft- tissue injury/contusion or strain; e.g. fracture, nerve injury, ligament disruption, tear of muscle or cartilage, or open wound
* current skin disorder or shaving hair at application site
* history of excessive sweating/hyperhidrosis inclusive of application site
* intake of non-steroidal anti-inflammatory drags (NSAIDs) or analgesics within 36 hours, opioids within 7 days, or corticosteroids (except inhaled corticosteroids for e.g. topical treatment of bronchial asthma) within 60 days of inclusion in the study
* intake of long-acting NSAIDs or application of topical medication since the injury (Rest, Ice, Compression, and elevation (RICE) allowed)
* participation in a clinical study within 30 days before inclusion in the study or concomitantly
* participation in this clinical study in another center
* drug or alcohol abuse in the opinion of the Investigator
* pregnant and lactating women
* women of child-bearing potential (defined as all women physiologically capable of becoming pregnant) who are not using an acceptable method of contraception defined as:

  * Surgical sterilization
  * Combined (estrogen and progestogen containing) hormonal contraception, e.g., oral, intravaginal, transdermal and progestogen-only hormonal contraception e.g. oral, injectable, implantable as well as intrauterine device (IUD) and intrauterine hormone-releasing system (IUS) each in combination with male condom to increase safety effect (double barrier method)
  * Total abstinence throughout the study at the discretion of the Investigator
  * Periodic abstinence is NOT an acceptable method of contraception. An acceptable method of contraception must be maintained throughout the study
  * A woman who is post-menopausal must have a negative urine pregnancy test at screening but will not need to comply with an acceptable method of contraception. Women are considered post-menopausal and not of child bearing potential if they had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of sterilisation, salpingectomy) or 6 months of spontaneous amenorrhea with serum Follic simulating hormone (FSH) levels > 40 mIU/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least 6 weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* known hypersensitivity to Esflurbiprofen, R-flurbiprofen or one of the excipients of the patch
* patients with any ongoing condition that may interfere with the absorption, distribution, metabolism, or excretion of Esflurbiprofen
* history of previous significant injury to the same extremity within 6 months
* patients with a disease affecting the same limb, such as synovitis, rheumatoid arthritis, arthrosis, etc.
* patients having an ongoing painful condition associated with blunt injury/contusion
* patients suffering from symptoms of an infectious disease including swelling of any joint of the affected lower limbs
* patients who had surgery of the affected lower limb within one year of study entry
* patients with significant diseases (defined as a disease which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study; includes patients with a history of gastrointestinal bleeding, significant cardiovascular, liver or renal disease)
* patients with a blood coagulation disorder
* patients who use any impermissible medication
* known allergy to paracetamol and galenic components of the rescue medication

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Sum of Pain Intensity Difference (SPID) on pain-on-movement (POM) over 0-48 hours | Day 1 to Day 3
  Calculating the area under the curve for the difference of each pain intensity score by 100-mm-Visual Analogue Scale (VAS) on movement from the baseline over 0-48 hours after patch application.

SECONDARY OUTCOMES:
100-mm- Visual Analogue Scale (VAS) score on pain-on-movement (POM) | Day 1 to Day 8
  VAS score from no pain (0 mm) to worst pain (100 mm) on pain-on-movement by a patient at each time point
100-mm- Visual Analogue Scale (VAS) score on pain-at-rest (PAR) | Day 1 to Day 8
  VAS score from no pain (0 mm) to worst pain (100 mm) on PAR (at least 5 min rest) by a patient at each time point
Sum of Pain Intensity Difference (SPID) on pain-on-movement (POM) | Day 1 to Day 8
  Calculating the area under the curve for the difference of each pain intensity score by 100-mm-Visual Analogue Scale (VAS) on movement from the baseline over day 1 to day 8.
Sum of Pain Intensity Difference (SPID) on pain-at-rest (PAR) | Day 1 to Day 8
  Calculating the area under the curve for the difference of each pain intensity score by 100-mm-Visual Analogue Scale (VAS) at rest from the baseline over day 1 to day 8.
Pain Intensity Difference (PID) on pain-on-movement (POM) | Day 1 to Day 8
  Difference of each pain intensity score by 100-mm-Visual Analogue Scale (VAS) on movement from the baseline at each time point.
Pain Intensity Difference (PID) on pain-at-rest (PAR) | Day 1 to Day 8
  Difference of each pain intensity score by 100-mm-Visual Analogue Scale (VAS) on movement from the baseline at each time point.
Time to meaningful/optimal reduction | Day 1 to Day 8
  Time to meaningful/optimal reduction of pain defined as first at least 30% (meaningful) and 50% (optimal) reduction from baseline of VAS on POM.
Time to complete resolution | Day 1 to Day 8
  * Time to complete resolution of POM VAS value of 0 mm
  * Time to complete resolution of PAR VAS value of 0 mm
Responder rate 1 | Day 3
  Responder rate is defined as the number of patients achieving at least 50% reduction from baseline in the VAS score for POM at 48 hours
Responder rate 2 | Day 8
  number of patients able to resume training / normal physical activity by 168 hours
Resolution of ankle sprain | Day 8
  the percentage of patients who showed POM=PAR=0 at 168 hours
Global efficacy assessments 1 by investigator | Day 3, Day 4 and Day 8
  The global efficacy assessments are evaluated by the Investigator as the response to following questions: "Considering how this treatment has affected the patient since he/she started in the study, how well is he/she doing?" It is assessed on the following 5-point Likert scale: 0 = very good, 1 = good, 2 = fair, 3 = poor, 4 = very poor
Global efficacy assessments 2 by investigator | Day 3, Day 4 and Day 8
  The global efficacy assessments are evaluated by the Investigator as the response to following questions: "How would you rate this medication for the treatment of this ankle sprain?" The evaluation is based on the following 5-point Likert scale: 0 = excellent, 1 = very good, 2 = good, 3 = moderate, 4 = poor
Global efficacy assessments 1 by patients | Day 3, Day 4 and Day 8
  The global efficacy assessments are evaluated by the Investigator as the response to following questions: "Considering how this treatment has affected you since you started in the study, how well are you doing?" It is assessed on the following 5-point Likert scale: 0 = very good, 1 = good, 2 = fair, 3 = poor, 4 = very poor
Global efficacy assessments 2 by patients | Day 3, Day 4 and Day 8
  The global efficacy assessments are evaluated by the patient as the response to following questions: "How do you rate this medication as a treatment for your ankle sprain?" It is assessed on the following 5-point Likert scale: 0 = excellent, 1 = very good, 2 = good, 3 = fair, 4 = poor
Number of use of rescue medication | Day 1 to Day 8
  Number of resucue medication use during clinical study
Number of patients who experience adverse event and serious adverse event | Day 1 to Day 8
  Characterization of occurrence of adverse events or serious adverse events of TK-254RX or placebo patch
Characterization of local tolerability | Day 8
  Assessing the local tolerability by using the 8-point dermal response (0: No evidence of irritation, 1: Minimal erythema, barely perceptible, 2: Definite erythema, readily visible, minimal edema or minimal papular response, 3: Erythema and papules, 4: Definite edema, 5: Erythema, edema, and papules, 6: Vesicular eruption, 7: Strong reaction spreading beyond test site) and other effects score (0: No other effect detected, A(0): Slightly glazed appearance, B(1): Markedly glazed appearance, C(2): Glazing with peeling and cracking, F(3): Glazing with fissures, G(3): Film of dried serous exudates covering all or part of the application site, H(3): Small petechial erosions and/or scabs) according to FDA recommendation
Patch adhesion assessed by the site staff | Day 2 to Day 5
  Adhesive power of the EFTS will be visually assessed and classified by the site staff in a 5-point-score (0=≥ 90% adhered / 1= ≥75% to <90% adhered / 2=≥50% to <75% adhered / 3=>0% to <50% adhered / 4=completely detached)
Patch adhesion assessed by patient | Day 1 to Day 8
  Adhesive power of the EFTS will be visually assessed and classified by a patient in a 5-point-score (0=≥ 90% adhered / 1= ≥75% to <90% adhered / 2=≥50% to <75% adhered / 3=>0% to <50% adhered / 4=completely detached)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Nishiyama, Study Chair — Teikoku Seiyaku Co., Ltd.
Locations (5):
- Germany (5):
  - Medical Practice Ebert, Siemensstr, Bonn
  - Medical Practice Prof. Predel, Siemensstr, Bonn
  - Medical Practice Schaale-Maas, Siemensstr, Bonn
  - Medical Practice Pabst, Sportschule Puch, Fürstenfeldbruck
  - Medical Practice Gastl, Römerstraße, Gilching

IPD SHARING:
Plan to Share IPD: No